CLINICAL TRIAL: NCT03788759
Title: Alpha-lipoic Acid Adjunctive Therapy in Schizophrenia: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Alpha-lipoic Acid Adjunctive Therapy in Schizophrenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nucleo De Pesquisa E Desenvolvimento De Medicamentos Da Universidade Federal Do Ceara (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Lia Sanders, Principal Investigator, Nucleo De Pesquisa E Desenvolvimento De Medicamentos Da Universidade Federal Do Ceara
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LipoicStudy
Record Dates: First submitted 2018-12-20; First posted 2018-12-28 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Schizophrenia; Oxidative Stress
Keywords: Schizophrenia; Drug repurposing; Alpha-lipoic acid; Adjuvant treatment
MeSH Terms: conditions — Schizophrenia | interventions — Thioctic Acid

STUDY DESIGN:
Intervention Model Description: Proof of concept 4-month prospective, randomized, double-blind, controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): 25 subjects will be randomized to 100mg of alpha-lipoic acid.
  Interventions: Drug: Alpha-lipoic acid
- Placebo group (Placebo Comparator): 25 subjects will be randomized to placebo.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Alpha-lipoic acid — Administration of ALA (100 mg/day) for 4 months, as an adjunct to antipsychotic medication.
  Arms: Experimental group
Drug: Placebo Oral Tablet — Administration of placebo, as an adjunct to antipsychotic medication.
  Arms: Placebo group

SUMMARY:
Schizophrenia is a devastating mental disorder with a prevalence of approximately 1% worldwide. While effective in reducing positive symptoms, current treatments have limited effects on cognitive and social cognition/processing deficits of schizophrenia, which are closely linked to real-world dysfunction and lack of socio-occupational integration. There is compelling evidence for impaired antioxidant defense system and inflammatory abnormalities in schizophrenia. A new therapeutic approach to the disease might well be to hinder oxidative damage, inflammation and its clinical sequelae. Alpha-lipoic acid (ALA) is a naturally occurring compound, synthesized in the mitochondria, that is currently approved to treat diabetic neuropathic pain. Drug repurposing is a fast, and cost-effective method that can overcome drug discovery challenges of targeting neuropsychiatric disorders. In a pilot investigation, adjunctive treatment with ALA led to robust improvement in negative and cognitive symptoms of ten patients with schizophrenia. This project aims to investigate the efficacy of ALA as a disease-modifying drug for the treatment of schizophrenia, by improving sociability and cognition, as well as to correlate patients' response with biomarkers that will shed light on the pathophysiology of this complex disease. It comprises 1) a prospective, randomized, double-blind, placebo-controlled trial to evaluate efficacy of ALA to treat cognitive and negative symptoms of patients with schizophrenia and 2) an investigation of changes in biomarkers of oxidative stress in response to adjunctive treatment with ALA. The proposed study could establish a new adjunctive treatment for schizophrenia, recognize a novel pharmacological approach and help unveil the biological basis of the disease.

DETAILED DESCRIPTION:
The underlying pathogenesis of schizophrenia remains unknown, but aberrant reduction-oxidation has gained increasing support as an hypothesis to help explain the pathophysiology of the disease. Alpha-lipoic acid (ALA) is a naturally occurring antioxidant, essential for the function of different enzymes of mitochondria's oxidative metabolism, that is currently approved to treat diabetic neuropathic pain9. ALA and its reduced form, dihydrolipoic acid (DHLA), have important advantages over other antioxidant agents such as vitamin E and C, partly due to their amphiphilic properties, which confer antioxidant actions in the membrane as well as in the cytosol. A preclinical study conducted in our lab showed that ALA alone and combined with clozapine reverses schizophrenia associated symptoms and pro-oxidant changes induced by ketamine in mice. Before the widespread use of antipsychotics, two studies found that low doses of ALA relieved symptoms in patients with schizophrenia.

More recently, my colleagues and I conducted an open label proof of concept study that provided encouraging evidence that low doses of ALA might be an effective adjunctive treatment for schizophrenia. Based on promising preliminary results, the investigators will now test ALA in a more rigorous placebo-controlled clinical study.

Specific Aim1: To conduct a prospective, randomized, double-blind, placebo-controlled trial to evaluate the efficacy of adjuvant treatment with low doses (100mg) of ALA to treat cognitive and negative symptoms of patients with schizophrenia. The investigators will randomize 50 patients over 4 months.

Specific Aim 2: To quantify changes in biomarkers of oxidative stress in response to adjunctive treatment with ALA. The hypothesis is that changes in these biomarkers will mediate the clinical response to ALA.

Research Plan: To carry out a proof of concept 4-month prospective, randomized, double-blind, controlled trial of alpha-lipoic acid, at doses of 100 mg/day or identical placebo tablets, added to ongoing antipsychotics in 50 stable patients (ages 18-60 years, 25 patients per group) with diagnosis of schizophrenia. The study will be conducted at the Drug Research and Development Center (NPDM), at the Universidade Federal do Ceará, Fortaleza, Brazil. This center has a long history of performing placebocontrolled trials in clinical medicine (http://www.npdm.ufc.br/) and has the necessary infrastructure to successfully complete the proposed study protocol. All participants will give written informed consent prior to study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to provide informed consent;
* Schizophrenia diagnosis (made by research psychiatrists using the Structured Clinical Interview, SCID-5, for Diagnostic and Statistical Manual of Mental Disorders);
* Negative and/or cognitive symptoms despite adequate antipsychotic treatment;
* Ages 18-60 years

Exclusion Criteria:

* 6-month history of any drug or alcohol abuse or dependence;
* Changes in psychotropic medications within the last 4 weeks;
* Actual valproate use (potential interaction with ALA);
* General medical illness including autoimmune disorders, known chronic infections such as HIV or hepatitis C, and liver or renal failure that could adversely impact on patient outcome;
* Women who are planning to become pregnant, are pregnant, or are breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change in the Brief Psychiatry Rating Scale (BPRS) scores | Baseline and 16 weeks
  18-item rating scale to assess changes in psychopathology; each item is scored 0-6, yielding a total between 0 and 108.

SECONDARY OUTCOMES:
Change in the Simpson-Angus Extrapyramidal Symptoms Scale (SAS) scores | Baseline and 16 weeks
  10-item rating scale to assess extrapyramidal symptoms; each item is scored 0-4, yielding a total between 0 and 40.
Brain resting state activity | Baseline and 16 weeks
  Functional Magnetic Resonance Imaging (fMRI) scans before and after treatment
Gut Microbiota Composition | Baseline and 16 weeks
  Analyses of patient's gut microbiota
Change in Body Mass Index (BMI) | Baseline and 16 weeks
  Weight and height will be combined to report BMI in kg/m^2
Change in Abdominal Circumference | Baseline and 16 weeks
  Abdominal Circumference in cm
Change in plasma Aspartate Aminotransferase (AST) | Baseline and 16 weeks
  AST in U/L
Change in plasma Aspartate Aminotransferase (AST) Alanine Aminotransferase (ALT) | Baseline and 16 weeks
  ALT in U/L
Change in Hemoglobin concentration (HC) | Baseline and 16 weeks
  HC in g/dL
Change in Hematocrit (Ht) | Baseline and 16 weeks
  Ht in %
Change in White blood cell count (WBC) | Baseline and 16 weeks
  WBC in number per microliter
Change in Neutrophil Count (NC) | Baseline and 16 weeks
  NC in number per microliter
Change in Platelet Count (PC) | Baseline and 16 weeks
  PC in number per microliter
Change in Glycohemoglobin (HbA1c) | Baseline and 16 weeks
  HbA1c in %
Change in serum level of Vitamin B12 | Baseline and 16 weeks
  Vitamin B12 in pg/mL
Change in serum level of Folic Acid | Baseline and 16 weeks
  Folic Acid in ng/mL
Change in Plasma Glutathione (GSH) | Baseline and 16 weeks
  GSH in ng/mL
Change in serum level of Nitrite | Baseline and 16 weeks
  Nitrite in nanomole/mililiter
Change in serum level of Thiobarbituric acid reactive substances (TBARS) | Baseline and 16 weeks
  TBARS in mmol of malonaldehyde/mL
Change in serum level of Interleukin 1 β (IL-1β) | Baseline and 16 weeks
  IL-1β in pg/mL
Change in serum level of Interleukin-4 | Baseline and 16 weeks
  IL-4 in pg/mL
Change in serum level of Interferon gamma (IFNγ) | Baseline and 16 weeks
  IFNγ in pg/mL
Change in serum level of Tumor necrosis factor alpha (TNF-α) | Baseline and 16 weeks
  TNF-α in pg/mL
Change in Indoleamine 2,3-dioxygenase (IDO) enzymatic activity | Baseline and 16 weeks
  IDO activity in U IDO mol^-1/mg^-1
Change in serum level of Eotaxin | Baseline and 16 weeks
  Eotaxin in ng/mL
Change in serum level of Isoprostanes | Baseline and 16 weeks
  Isoprostanes in pg/mL
Change in serum level of Calprotectin | Baseline and 16 weeks
  Serum Calprotectin in ng/mL
Change in serum level of Serotonin | Baseline and 16 weeks
  Serotonin in ng/mL
Change in Block Corsi Test | Baseline and 16 weeks
  This test assesses visuo-spatial short term working memory. Participants are asked to mimick a researcher as he/she taps a sequence of up to nine identical spatially separated blocks. The test measures both the number of correct sequences and the longest sequence remembered.
Change in serum level of Tryptophan | Baseline and 16 weeks
  Tryptophan in micrograms/mL
Change in Trail Making Test | Baseline and 16 weeks
  Trail Making Test measured in time and number of errors. It tests visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. Provide information about visual search speed, scanning, speed of processing, mental flexibility, executive functioning.
Change in Subtest Digit Span | Baseline and 16 weeks
  Individual tries to repeat digits forward, backward, and in ascending order. This test measures short term memory, working memory. The score is the maximum number of digits correctly remembered.
Category (Animal) Fluency | Baseline and 16 weeks
  Participants have to produce as many words as possible from a category in a given time (usually 60 seconds). Performance measure is the total number of words
F-A-S test | Baseline and 16 weeks
  It assesses phonemic fluency by requesting an individual to orally produce as many words as possible that begin with the letters F, A, and S within a prescribed time frame, usually 1 min.
Rey Auditory Verbal Learning Test | Baseline and 16 weeks
  Participants are asked to repeat list of 15 unrelated words; another list of 15 unrelated words are given and participants must again repeat the original list of 15 words and then again after 30 minutes. Score range: 0-15

CONTACTS AND LOCATIONS:
Overall Officials: Lia LO Sanders, MD, PhD, Principal Investigator — Núcleo de Pesquisa e Desenvolvimento de Medicamentos
Locations (1):
- Núcleo de Pesquisa e Desenvolvimento de Medicamentos - UFC, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Perala J, Suvisaari J, Saarni SI, Kuoppasalmi K, Isometsa E, Pirkola S, Partonen T, Tuulio-Henriksson A, Hintikka J, Kieseppa T, Harkanen T, Koskinen S, Lonnqvist J. Lifetime prevalence of psychotic and bipolar I disorders in a general population. Arch Gen Psychiatry. 2007 Jan;64(1):19-28. doi: 10.1001/archpsyc.64.1.19. PMID 17199051
- [Background] Foussias G, Agid O, Fervaha G, Remington G. Negative symptoms of schizophrenia: clinical features, relevance to real world functioning and specificity versus other CNS disorders. Eur Neuropsychopharmacol. 2014 May;24(5):693-709. doi: 10.1016/j.euroneuro.2013.10.017. Epub 2013 Nov 11. PMID 24275699
- [Background] Reddy RD, Yao JK. Free radical pathology in schizophrenia: a review. Prostaglandins Leukot Essent Fatty Acids. 1996 Aug;55(1-2):33-43. doi: 10.1016/s0952-3278(96)90143-x. PMID 8888121
- [Background] Bitanihirwe BK, Woo TU. Oxidative stress in schizophrenia: an integrated approach. Neurosci Biobehav Rev. 2011 Jan;35(3):878-93. doi: 10.1016/j.neubiorev.2010.10.008. Epub 2010 Oct 23. PMID 20974172
- [Background] Gysin R, Kraftsik R, Boulat O, Bovet P, Conus P, Comte-Krieger E, Polari A, Steullet P, Preisig M, Teichmann T, Cuenod M, Do KQ. Genetic dysregulation of glutathione synthesis predicts alteration of plasma thiol redox status in schizophrenia. Antioxid Redox Signal. 2011 Oct 1;15(7):2003-10. doi: 10.1089/ars.2010.3463. Epub 2010 Oct 30. PMID 20673128
- [Background] Fournier M, Ferrari C, Baumann PS, Polari A, Monin A, Bellier-Teichmann T, Wulff J, Pappan KL, Cuenod M, Conus P, Do KQ. Impaired metabolic reactivity to oxidative stress in early psychosis patients. Schizophr Bull. 2014 Sep;40(5):973-83. doi: 10.1093/schbul/sbu053. Epub 2014 Mar 31. PMID 24687046
- [Background] Prabakaran S, Swatton JE, Ryan MM, Huffaker SJ, Huang JT, Griffin JL, Wayland M, Freeman T, Dudbridge F, Lilley KS, Karp NA, Hester S, Tkachev D, Mimmack ML, Yolken RH, Webster MJ, Torrey EF, Bahn S. Mitochondrial dysfunction in schizophrenia: evidence for compromised brain metabolism and oxidative stress. Mol Psychiatry. 2004 Jul;9(7):684-97, 643. doi: 10.1038/sj.mp.4001511. PMID 15098003
- [Background] Vallianou N, Evangelopoulos A, Koutalas P. Alpha-lipoic Acid and diabetic neuropathy. Rev Diabet Stud. 2009 Winter;6(4):230-6. doi: 10.1900/RDS.2009.6.230. Epub 2009 Dec 30. PMID 20043035
- [Background] Scott BC, Aruoma OI, Evans PJ, O'Neill C, Van der Vliet A, Cross CE, Tritschler H, Halliwell B. Lipoic and dihydrolipoic acids as antioxidants. A critical evaluation. Free Radic Res. 1994 Feb;20(2):119-33. doi: 10.3109/10715769409147509. PMID 7516789
- [Background] Vasconcelos GS, Ximenes NC, de Sousa CN, Oliveira Tde Q, Lima LL, de Lucena DF, Gama CS, Macedo D, Vasconcelos SM. Alpha-lipoic acid alone and combined with clozapine reverses schizophrenia-like symptoms induced by ketamine in mice: Participation of antioxidant, nitrergic and neurotrophic mechanisms. Schizophr Res. 2015 Jul;165(2-3):163-70. doi: 10.1016/j.schres.2015.04.017. Epub 2015 Apr 30. PMID 25937462
- [Background] GIAMATTEI L. [Thioctic acid in therapy of schizophrenia]. Osp Psichiatr. 1957 Apr-Jun;25(2):221-8. No abstract available. Italian. PMID 13526963
- [Background] ALTSCHULE MD, GONCZ RM, HOLLIDAY PD. Carbohydrate metabolism in brain disease. XI. Effects of thioctic (alpha-lipoic) acid in chronic schizophrenia. AMA Arch Intern Med. 1959 May;103(5):726-9. doi: 10.1001/archinte.1959.00270050048008. No abstract available. PMID 13636491
- [Background] Emsley R, Chiliza B, Asmal L, du Plessis S, Phahladira L, van Niekerk E, van Rensburg SJ, Harvey BH. A randomized, controlled trial of omega-3 fatty acids plus an antioxidant for relapse prevention after antipsychotic discontinuation in first-episode schizophrenia. Schizophr Res. 2014 Sep;158(1-3):230-5. doi: 10.1016/j.schres.2014.06.004. Epub 2014 Jul 2. PMID 24996507
- [Background] Kim E, Park DW, Choi SH, Kim JJ, Cho HS. A preliminary investigation of alpha-lipoic acid treatment of antipsychotic drug-induced weight gain in patients with schizophrenia. J Clin Psychopharmacol. 2008 Apr;28(2):138-46. doi: 10.1097/JCP.0b013e31816777f7. PMID 18344723
- [Background] Seybolt SE. Less is more. Schizophr Res. 2014 Dec;160(1-3):222-3. doi: 10.1016/j.schres.2014.10.022. Epub 2014 Oct 31. No abstract available. PMID 25458573
- [Background] Sanders LLO, de Souza Menezes CE, Chaves Filho AJM, de Almeida Viana G, Fechine FV, Rodrigues de Queiroz MG, Goncalvez da Cruz Fonseca S, Mendes Vasconcelos SM, Amaral de Moraes ME, Gama CS, Seybolt S, de Moura Campos E, Macedo D, Freitas de Lucena D. alpha-Lipoic Acid as Adjunctive Treatment for Schizophrenia: An Open-Label Trial. J Clin Psychopharmacol. 2017 Dec;37(6):697-701. doi: 10.1097/JCP.0000000000000800. PMID 29053478
- [Background] Steibliene V, Bunevicius A, Savickas A, Prange AJ Jr, Nemeroff CB, Bunevicius R. Triiodothyronine accelerates and enhances the antipsychotic effect of risperidone in acute schizophrenia. J Psychiatr Res. 2016 Feb;73:9-16. doi: 10.1016/j.jpsychires.2015.11.007. Epub 2015 Dec 1. PMID 26679760
- [Background] Ying Z, Kampfrath T, Sun Q, Parthasarathy S, Rajagopalan S. Evidence that alpha-lipoic acid inhibits NF-kappaB activation independent of its antioxidant function. Inflamm Res. 2011 Mar;60(3):219-25. doi: 10.1007/s00011-010-0256-7. Epub 2010 Oct 7. PMID 20927568
- [Background] Sola S, Mir MQ, Cheema FA, Khan-Merchant N, Menon RG, Parthasarathy S, Khan BV. Irbesartan and lipoic acid improve endothelial function and reduce markers of inflammation in the metabolic syndrome: results of the Irbesartan and Lipoic Acid in Endothelial Dysfunction (ISLAND) study. Circulation. 2005 Jan 25;111(3):343-8. doi: 10.1161/01.CIR.0000153272.48711.B9. Epub 2005 Jan 17. PMID 15655130
- [Background] Kanchanatawan B, Hemrungrojn S, Thika S, Sirivichayakul S, Ruxrungtham K, Carvalho AF, Geffard M, Anderson G, Maes M. Changes in Tryptophan Catabolite (TRYCAT) Pathway Patterning Are Associated with Mild Impairments in Declarative Memory in Schizophrenia and Deficits in Semantic and Episodic Memory Coupled with Increased False-Memory Creation in Deficit Schizophrenia. Mol Neurobiol. 2018 Jun;55(6):5184-5201. doi: 10.1007/s12035-017-0751-8. Epub 2017 Sep 5. PMID 28875464
- [Derived] Frota IJ, de Oliveira ALB, De Lima DN Jr, Costa Filho CWL, Menezes CES, Soares MVR, Chaves Filho AJM, Los DB, Moreira RTA, Viana GA, Campos EM, Vasconcelos SMM, Seeman MV, Macedo DS, Sanders LLO. Decrease in cognitive performance and increase of the neutrophil-to-lymphocyte and platelet-to-lymphocyte ratios with higher doses of antipsychotics in women with schizophrenia: a cross-sectional study. BMC Psychiatry. 2023 Aug 2;23(1):558. doi: 10.1186/s12888-023-05050-x. PMID 37532985
- [Derived] De Lima DN Jr, Costa Filho CWL, Frota IJ, de Oliveira ALB, Menezes CES, Chaves Filho AJM, Viana GA, Campos EM, Collares M, de Queiroz MGR, da Cruz Fonseca SG, Vasconcelos SMM, Macedo DS, Sanders LLO. alpha-Lipoic Acid as Adjunctive Treatment for Schizophrenia: A Randomized Double-Blind Study. J Clin Psychopharmacol. 2023 Jan-Feb 01;43(1):39-45. doi: 10.1097/JCP.0000000000001639. PMID 36584248